CLINICAL TRIAL: NCT04285827
Title: A 2-Part, Phase 1, Multi-Center, Single-Dose, Open Label, Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of CSL889 in Adult Patients With Sickle Cell Disease
Brief Title: Safety of Single Doses of CSL889 in Adult Patients With Sickle Cell Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CSL889_1001; 2019-001870-27 (EudraCT Number)
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- CSL889 Cohort A1 (Dose 1) (Experimental): CSL889 administered as a single IV infusion
  Interventions: Biological: CSL889
- CSL889 Cohort A2 (Dose 2) (Experimental): CSL889 administered as a single IV infusion
  Interventions: Biological: CSL889
- CSL889 Cohort A3 (Dose 3) (Experimental): CSL889 administered as a single IV infusion
  Interventions: Biological: CSL889
- CSL889 Cohort A4 (Dose 4) (Experimental): CSL889 administered as a single IV infusion
  Interventions: Biological: CSL889
- CSL889 Cohort A5 (Dose 5) (Experimental): CSL889 administered as a single IV infusion
  Interventions: Biological: CSL889
- CSL889 Cohort A6 (Dose 6) (Experimental): CSL889 administered as a single IV infusion
  Interventions: Biological: CSL889
- CSL889 Cohort B1 (low dose) (Experimental): CSL889 administered as a single IV infusion
  Interventions: Biological: CSL889
- CSL889 Cohort B2 (high dose) (Experimental): CSL889 administered as a single IV infusion
  Interventions: Biological: CSL889

INTERVENTIONS:
Biological: CSL889 — Administered as an IV infusion

SUMMARY:
This is a phase 1, first-in-human, multi-center, open-label, single dose cohort study to evaluate the safety and tolerability, pharmacokinetics (PK), exploratory pharmacodynamics (PD), and biomarkers of target engagement of CSL889 following single intravenous (IV) doses in subjects with sickle cell disease (SCD). The study involves sequential dose escalation of cohorts with between-group assessments of key safety and PK variables.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SCD as documented in the subject's medical record
* Aged 18 to 60 years, inclusive
* Stable SCD for at least 30 days before Day 1. Stable SCD is defined as the subject being at his or her medical baseline, with no evidence of worsening of disease over the last 30 days (including VOC, recent major surgery, hospitalization, serious infection, significant bleeding, cerebrovascular accident, seizures, or IV opioids)(Part A)
* Uncomplicated VOC requiring parenteral opioid treatment and admission to hospital for management. Uncomplicated VOC is defined as sickle cell pain without the following associated clinical features (Part B):

  * Fever (> 38.5 °C)
  * Hypotension (< 90/60 mmHg)
  * Hypoxia (< 90% oxygen saturation on room air, or requiring oxygen therapy to maintain oxygen saturation above 90%)
  * New neurological signs and / or symptoms clinically suggestive of stroke or transient ischemic attack
  * Signs and / or symptoms of Acute Chest Syndrome, accompanied by any new pulmonary infiltrate on chest radiography (chest X-ray to be performed if clinically indicated and according to local clinical guidelines)
* Subject is either not taking one of the study permitted SCD therapies (hydroxyurea, L-glutamine, L-glutaminecrizanlizumab, and/or voxelotor) or subject has been taking one or more of those for at least 30 days before Day 1 and is on a stable, well tolerated regimen that is planned to continue without change throughout the study

Exclusion Criteria:

* History of primary hemorrhagic stroke
* History or evidence of inherited bleeding diathesis or significant coagulopathy at risk for bleeding
* Weight >110 kg (242 lbs)
* Surgery within 30 days before Day 1 or any preplanned surgeries during the study (minor surgeries may be permitted under local anesthesia before screening, with permission of the medical monitor)
* Female subjects who are pregnant or breastfeeding
* Female subject of childbearing potential or fertile male subject either not using or not willing to use an acceptable method of contraception to avoid pregnancy during the study and for 30 days after receipt of CSL889.
* Treatment with any other drug / biologic that is newly approved for SCD during the conduct of this study within 90 days before Day 1. Exceptions: crizanlizumab [Adakveo®] and voxelotor [Oxbryta®] ] are permitted (where prescribed).
* Treatment with another investigational product within 30 days or within 5 half-lives of the product (whichever is greater) before Day 1
* Vaccination within 30 days before Day 1, or planned vaccination during the study
* Body-mass index < 16 kg/m2 or weight < 50 kg (110 lbs)
* History of anaphylactic-type reactions, transfusion related reaction, asthma, or autoimmune disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with treatment-emergent adverse events (TEAEs) by Cohort | Up to 32 days after start of CSL889 infusion
Percentage of subjects with TEAEs by severity by Cohort | Up to 32 days after start of CSL889 infusion
Percentage of subjects with TEAEs by causality by Cohort | Up to 32 days after start of CSL889 infusion

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) of CSL889 by Cohort | Up to 32 days after CSL889 infusion
Area under CSL889 serum concentration-time curve (AUC) from time 0 to time t (AUC0-t) by Cohort | Up to 32 days after CSL889 infusion
Maximum observed serum concentration (Cmax) of CSL889 by Cohort AUC extrapolated to infinity (AUC0-inf) by CSL889 dose level | Up to 32 days after CSL889 infusion
Time of Cmax (tmax) of CSL889 by Cohort | Up to 32 days after CSL889 infusion
Terminal half-life (t1/2) of CSL889 by Cohort | Up to 32 days after CSL889 infusion
Clearance (CL) of CSL889 by Cohort | Up to 32 days after CSL889 infusion
Volume of distribution (Vz) of CSL889 by Cohort | Up to 32 days after CSL889 infusion
Percentage of subjects with detectable antibodies to CSL889 by Cohort | Up to 32 days after CSL889 infusion

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (15):
- United States (8):
  - University of Illinois Hospital and Health Science Systems, Chicago, Illinois
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Jacobi Medical Center, The Bronx, New York
  - Brody School of Medicine at East Carolina University, Greenville, North Carolina
  - Ohio State University, Columbus, Ohio
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
- Netherlands (2):
  - Amsterdam UMC Academic Medical Center, Amsterdam
  - Erasmus University Medical Center, Rotterdam
- United Kingdom (5):
  - Liverpool University Hospital, Liverpool
  - Guys and St. Thomas, London
  - University College London Hospital, London
  - Manchester University Hospitals NHS Foundation Trust / Manchester Royal Infirmary, Manchester
  - Early Phase Unit, Manchester

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider requests to share Individual Patient Data (IPD) from systematic review groups or bona-fide researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.
Supporting Information: Study Protocol, SAP
Time Frame: IPD requests may be submitted to CSL no earlier than 12 months after publication of the results of this study via an article made available on a public website.
Access Criteria: Requests may only be made by systematic review groups or bona-fide researchers whose proposed use of the IPD is non-commercial in nature and has been approved by an internal review committee.
  An IPD request will not be considered by CSL unless the proposed research question seeks to answer a significant and unknown medical science or patient care question as determined by CSL's internal review committee.
  The requesting party must execute an appropriate data sharing agreement before IPD will be made available.